CLINICAL TRIAL: NCT01077856
Title: GARDASIL™ Vaccine Impact in Population Study
Brief Title: GARDASIL™ Vaccine Impact in Population Study (V501-033)
Acronym: VIP
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Danish Cancer Society (Other); Union for International Cancer Control (Other); Norwegian Institute of Public Health (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: V501-033; 2010_018 (Other: Merck Registration Number); EP08014.033 (Other: Merck Study Number)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Human Papillomavirus Infections
Keywords: congenital anomaly; pregnancy; GARDASIL®; Nordic; population-based
MeSH Terms: conditions — Papillomavirus Infections; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tissue, cervical cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pre-Vaccine: Registry, survey, and HPV status data from 2004-2006
- Post-Vaccine: Registry, survey, and HPV status data from 2011-2012

SUMMARY:
This study will assess the impact of GARDASIL™ human papillomavirus (HPV) vaccine in the general female population by utilizing nationwide registry databases in the participating Nordic countries.

DETAILED DESCRIPTION:
Time perspective: The study will be conducted using data collected both retrospectively/concurrently from registries and prospectively by questionnaire survey.

Baseline survey data were collected during a prior study from 2004-2005.

Safety Monitoring: An expert panel on teratology consisting of one teratologist from each of the participating countries will review all available medical records related to any congenital anomalies to search for any emerging patterns that may be indicative of an association between GARDASIL™ exposure in the mother and the subsequent congenital anomalies in the babies.

ELIGIBILITY:
Inclusion Criteria: - Registry Data: * Female residents of participating Nordic countries who were alive on January 1st in the year the data will be used for analysis - Survey Data: --Female residents alive in the participating countries on July 1, 2011 --Women must provide consent to use questionnaire data and to link data to other registry databases - Cervical Sample Collection: --For HPV data in the general population: cervical samples from residents of the participating countries who are 45 years and under collected between 2006 and 2007, or in 2011-2012 --For HPV data in lesional samples: cervical samples from women with a diagnosis of CIN or cervical cancer between 2004-2006 and 2011-2012 Exclusion Criteria: - Registry Data: * Women who participated in Protocol V501-015 (NCT00092534) and are included in the Long-Term Follow-Up study - Survey Data: --Women under 18 or above age 45 on July 1, 2011 --Women who participated in Protocol V501-015 and are included in the Long-Term Follow-Up study - Cervical Sample Collection: --Samples from women who participated in Protocol V501-015 and are included in the Long-Term Follow-Up study --Samples with inadequate integrity for HPV testing

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Registry data from the Population, Cervical Cancer Screening, Pathology, Cancer, and Death registries; Survey: Questionnaire sent to random sampling of women from the Central Population Registry Database; HPV Data: liquid-based cytology and histology samples from hospitals in participating countries
Sampling Method: Probability Sample
Enrollment: 54516 (Actual)
Dates: Start 2007-05-29 (Actual); Primary Completion 2014-12-02 (Actual); Study Completion 2014-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Bonanni P, Cohet C, Kjaer SK, Latham NB, Lambert PH, Reisinger K, Haupt RM. A summary of the post-licensure surveillance initiatives for GARDASIL/SILGARD. Vaccine. 2010 Jul 5;28(30):4719-30. doi: 10.1016/j.vaccine.2010.04.070. Epub 2010 May 6. PMID 20451636
- [Result] Baldur-Felskov B, Dehlendorff C, Munk C, Kjaer SK. Early impact of human papillomavirus vaccination on cervical neoplasia--nationwide follow-up of young Danish women. J Natl Cancer Inst. 2014 Mar;106(3):djt460. doi: 10.1093/jnci/djt460. Epub 2014 Feb 19. PMID 24552678
- [Derived] Nygard M, Hansen BT, Kjaer SK, Hortlund M, Tryggvadottir L, Munk C, Lagheden C, Sigurdardottir LG, Campbell S, Liaw KL, Dillner J. Human papillomavirus genotype-specific risks for cervical intraepithelial lesions. Hum Vaccin Immunother. 2021 Apr 3;17(4):972-981. doi: 10.1080/21645515.2020.1814097. Epub 2020 Sep 29. PMID 32990181
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V501-033&kw=V501-033&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Denmark Participants: Participants in Denmark who completed the first survey (before licensure of GARDASIL)
- Norway Participants: Participants in Norway who completed the first survey (before licensure of GARDASIL)
- Sweden Participants: Participants in Sweden who completed the first survey (before licensure of GARDASIL)
Period: Overall Study
Arm/Group | Denmark Participants | Norway Participants | Sweden Participants
Started | 22199 | 16604 | 15713
Completed | 22199 | 16604 | 15713
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who took the first survey given before Gardasil licensure
Groups:
- Total: Total of all reporting groups
Arm/Group | Denmark Participants | Norway Participants | Sweden Participants | Total
Number analyzed (Participants) | 22199 | 16604 | 15713 | 54516
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 31.9 [24.3 to 39.0] | 31.0 [24.0 to 38.0] | 33.2 [26.1 to 39.5] | 32.0 [24.8 to 39.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22199 | 16604 | 15713 | 54516
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Histologically-confirmed Cervical Intraepithelial Neoplasia (CIN) for Participants of All Ages in Denmark
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. The collection of such data in these registries is mandated by law and compliance is generally very high. The number of new cases of high-grade (2/3) CIN registered during the assessment periods in Denmark was recorded. Incidence rates are for all age groups and were age-adjusted using the European Standard Population. The incidence before Gardasil licensure is an average over the 3-year period.
Time Frame: Three years before Gardasil licensure (2004 to 2006 combined) and annually after Gardasil licensure (2007, 2008, 2009, 2010, and 2011)
Population: The analysis population was the entire population of qualifying women in Denmark and thus changed throughout the analysis. The number of participants analyzed given below is an estimate calculated from the number of reported cases and the incidence data.
Measure: Number; unit: Cases per 100,000 women
Units Other Than Participants: cases
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2007, After Gardasil Licensure | Denmark Participants 2008 After Gardasil Licensure | Denmark Participants 2009 After Gardasil Licensure | Denmark Participants 2010 After Gardasil Licensure | Denmark Participants 2011 After Gardasil Licensure
Number analyzed (Participants) | 2531060 | 2521944 | 2509417 | 2513941 | 2504258 | 2495192
Number analyzed (cases) | 4156 | 4827 | 5463 | 6041 | 5587 | 5709
Cases per 100,000 women | 164.2 | 191.4 | 217.7 | 240.3 | 223.1 | 228.8

2. Primary Outcome: Incidence of Histologically-confirmed Cervical Intraepithelial Neoplasia for Participants <=26 Years of Age in Denmark
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. The collection of such data in these registries is mandated by law and compliance is generally very high. The number of new cases of high-grade (2/3) CIN registered during the assessment periods in Denmark was recorded. Incidence rates are for women <=26 years of age and were age-adjusted using the European Standard Population. The incidence before Gardasil licensure is an average over the 3-year period.
Time Frame: as for outcome 1
Population: The analysis population was the entire population of qualifying women <=26 years of age in Denmark and thus changed throughout the analysis. The number of participants analyzed given below is an estimate calculated from the number of reported cases and the incidence data.
Measure: Number; unit: Cases per 100,000 women
Units Other Than Participants: cases
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2007, After Gardasil Licensure | Denmark Participants 2008 After Gardasil Licensure | Denmark Participants 2009 After Gardasil Licensure | Denmark Participants 2010 After Gardasil Licensure | Denmark Participants 2011 After Gardasil Licensure
Number analyzed (Participants) | 711394 | 706535 | 700886 | 708048 | 873445 | 898759
Number analyzed (cases) | 949 | 1146 | 1345 | 1654 | 1615 | 1811
Cases per 100,000 women | 133.4 | 162.2 | 191.9 | 233.6 | 184.9 | 201.5

3. Primary Outcome: Incidence of Histologically-confirmed Cervical Intraepithelial Neoplasia for Participants >26 Years of Age in Denmark
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. The collection of such data in these registries is mandated by law and compliance is generally very high. The number of new cases of high-grade (2/3) CIN registered during the assessment periods in Denmark was recorded. Incidence rates are for women >26 years of age and were age-adjusted using the European Standard Population. The incidence before Gardasil licensure is an average over the 3-year period.
Time Frame: as for outcome 1
Population: The analysis population was the entire population of qualifying women >26 years of age in Denmark and thus changed throughout the analysis. The number of participants analyzed given below is an estimate calculated from the number of reported cases and the incidence data.
Measure: Number; unit: Cases per 100,000 women
Units Other Than Participants: cases
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2007, After Gardasil Licensure | Denmark Participants 2008 After Gardasil Licensure | Denmark Participants 2009 After Gardasil Licensure | Denmark Participants 2010 After Gardasil Licensure | Denmark Participants 2011 After Gardasil Licensure
Number analyzed (Participants) | 1786630 | 1786893 | 1785776 | 1798688 | 1606146 | 1583909
Number analyzed (cases) | 3207 | 3681 | 4118 | 4387 | 3972 | 3898
Cases per 100,000 women | 179.5 | 206.0 | 230.6 | 243.9 | 247.3 | 246.1

4. Primary Outcome: Incidence of Histologically-confirmed Cervical Intraepithelial Neoplasia for Participants of All Ages in Norway
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. The collection of such data in these registries is mandated by law and compliance is generally very high. The number of new cases of high-grade (2/3) CIN registered during the assessment periods in Norway was recorded. Incidence rates are for all age groups and were age-adjusted using the European Standard Population. The incidence before Gardasil licensure is an average over the 3-year period.
Time Frame: as for outcome 1
Population: The analysis population was the entire population of qualifying women in Norway and thus changed throughout the analysis. The number of participants analyzed given below is an estimate calculated from the number of reported cases and the incidence data.
Measure: Number; unit: Cases per 100,000 women
Units Other Than Participants: cases
Arm/Group | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2007, After Gardasil Licensure | Norway Participants 2008 After Gardasil Licensure | Norway Participants 2009 After Gardasil Licensure | Norway Participants 2010 After Gardasil Licensure | Norway Participants 2011 After Gardasil Licensure
Number analyzed (Participants) | 2255064 | 2265583 | 2279310 | 2302533 | 2323589 | 2353224
Number analyzed (cases) | 3006 | 3344 | 3305 | 3364 | 3418 | 3431
Cases per 100,000 women | 133.3 | 147.6 | 145.0 | 146.1 | 147.1 | 145.8

5. Primary Outcome: Incidence of Histologically-confirmed Cervical Intraepithelial Neoplasia for Participants <=26 Years of Age in Norway
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. The collection of such data in these registries is mandated by law and compliance is generally very high. The number of new cases of high-grade (2/3) CIN registered during the assessment periods in Norway was recorded. Incidence rates are for women <=26 years of age and were age-adjusted using the European Standard Population. The incidence before Gardasil licensure is an average over the 3-year period.
Time Frame: as for outcome 1
Population: The analysis population was the entire population of qualifying women <=26 years of age in Norway and thus changed throughout the analysis. The number of participants analyzed given below is an estimate calculated from the number of reported cases and the incidence data.
Measure: Number; unit: Cases per 100,000 women
Units Other Than Participants: cases
Arm/Group | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2007, After Gardasil Licensure | Norway Participants 2008 After Gardasil Licensure | Norway Participants 2009 After Gardasil Licensure | Norway Participants 2010 After Gardasil Licensure | Norway Participants 2011 After Gardasil Licensure
Number analyzed (Participants) | 761571 | 773333 | 788991 | 806268 | 825000 | 854137
Number analyzed (cases) | 543 | 580 | 516 | 566 | 627 | 609
Cases per 100,000 women | 71.3 | 75.0 | 65.4 | 70.2 | 76.0 | 71.3

6. Primary Outcome: Incidence of Histologically-confirmed Cervical Intraepithelial Neoplasia for Participants >26 Years of Age in Norway
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. The collection of such data in these registries is mandated by law and compliance is generally very high. The number of new cases of high-grade (2/3) CIN registered during the assessment periods in Norway was recorded. Incidence rates are for women >26 years of age were age-adjusted using the European Standard Population. The incidence before Gardasil licensure is an average over the 3-year period.
Time Frame: as for outcome 1
Population: The analysis population was the entire population of women >26 years of age in Norway and thus changed throughout the analysis. The number of participants analyzed given below is an estimate calculated from the number of reported cases and the incidence data.
Measure: Number; unit: Cases per 100,000 women
Units Other Than Participants: cases
Arm/Group | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2007, After Gardasil Licensure | Norway Participants 2008 After Gardasil Licensure | Norway Participants 2009 After Gardasil Licensure | Norway Participants 2010 After Gardasil Licensure | Norway Participants 2011 After Gardasil Licensure
Number analyzed (Participants) | 1426999 | 1426949 | 1427329 | 1440783 | 1451378 | 1462176
Number analyzed (cases) | 2463 | 2764 | 2789 | 2798 | 2791 | 2822
Cases per 100,000 women | 172.6 | 193.7 | 195.4 | 194.2 | 192.3 | 193.0

7. Primary Outcome: Incidence of Histologically-confirmed Cervical Intraepithelial Neoplasia for Participants of All Ages in Sweden
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. The collection of such data in these registries is mandated by law and compliance is generally very high. The number of new cases of high-grade (2/3) CIN registered during the assessment periods in Sweden was recorded. Incidence rates are for all age groups and were age-adjusted using the European Standard Population. The incidence before Gardasil licensure is an average over the 3-year period.
Time Frame: as for outcome 1
Population: The analysis population was the entire population of qualifying women in Sweden and thus changed throughout the analysis. The number of participants analyzed given below is an estimate calculated from the number of reported cases and the incidence data.
Measure: Number; unit: Cases per 100,000 women
Units Other Than Participants: cases
Arm/Group | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2007, After Gardasil Licensure | Sweden Participants 2008 After Gardasil Licensure | Sweden Participants 2009 After Gardasil Licensure | Sweden Participants 2010 After Gardasil Licensure | Sweden Participants 2011 After Gardasil Licensure
Number analyzed (Participants) | 4187237 | 4188266 | 4199295 | 4243293 | 4432481 | 4357284
Number analyzed (cases) | 5971 | 6496 | 7143 | 6959 | 7451 | 8793
Cases per 100,000 women | 142.6 | 155.1 | 170.1 | 164.0 | 168.1 | 201.8

8. Primary Outcome: Incidence of Histologically-confirmed Cervical Intraepithelial Neoplasia for Participants <=26 Years of Age in Sweden
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. The collection of such data in these registries is mandated by law and compliance is generally very high. The number of new cases of high-grade (2/3) CIN registered during the assessment periods in Sweden was recorded. Incidence rates are for women <=26 years of age and were age-adjusted using the European Standard Population. The incidence before Gardasil licensure is an average over the 3-year period.
Time Frame: as for outcome 1
Population: The analysis population was the entire population of qualifying women <=26 years of age in Sweden and thus changed throughout the analysis. The number of participants analyzed given below is an estimate calculated from the number of reported cases and the incidence data.
Measure: Number; unit: Cases per 100,000 women
Units Other Than Participants: cases
Arm/Group | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2007, After Gardasil Licensure | Sweden Participants 2008 After Gardasil Licensure | Sweden Participants 2009 After Gardasil Licensure | Sweden Participants 2010 After Gardasil Licensure | Sweden Participants 2011 After Gardasil Licensure
Number analyzed (Participants) | 1461211 | 1462312 | 1548040 | 1605284 | 1672941 | 1724747
Number analyzed (cases) | 1375 | 1455 | 2014 | 2005 | 2133 | 2732
Cases per 100,000 women | 94.1 | 99.5 | 130.1 | 124.9 | 127.5 | 158.4

9. Primary Outcome: Incidence of Histologically-confirmed Cervical Intraepithelial Neoplasia for Participants >26 Years of Age in Sweden
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. The collection of such data in these registries is mandated by law and compliance is generally very high. The number of new cases of high-grade (2/3) CIN registered during the assessment periods in Sweden was recorded. Incidence rates are for women >26 years of age and were age-adjusted using the European Standard Population. The incidence before Gardasil licensure is an average over the 3-year period.
Time Frame: as for outcome 1
Population: The analysis population was the entire population of qualifying women >26 years of age in Sweden and thus changed throughout the analysis. The number of participants analyzed given below is an estimate calculated from the number of reported cases and the incidence data.
Measure: Number; unit: Cases per 100,000 women
Units Other Than Participants: cases
Arm/Group | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2007, After Gardasil Licensure | Sweden Participants 2008 After Gardasil Licensure | Sweden Participants 2009 After Gardasil Licensure | Sweden Participants 2010 After Gardasil Licensure | Sweden Participants 2011 After Gardasil Licensure
Number analyzed (Participants) | 3264205 | 3262783 | 2628908 | 2627821 | 2639206 | 2642110
Number analyzed (cases) | 4596 | 5041 | 5129 | 4945 | 5318 | 6061
Cases per 100,000 women | 140.8 | 154.5 | 195.1 | 188.1 | 201.5 | 229.4

10. Primary Outcome: Incidence of Human Papillomavirus (HPV) 6/11/16/18-related Cervical Intraepithelial Neoplasia for Participants of All Ages
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. In addition, lesional tissue samples were routinely collected and stored; the 2004 to 2006 period was chosen because it was sufficiently recent to reflect HPV type status immediately before licensure of Gardasil. The number of new cases of HPV 6/11/16/18-related high-grade (2/3) CIN was estimated based on the proportion of HPV 6/11/16/18 in all CIN in a representative sample. Incidence was age-adjusted according to Nordic Standard Population.
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: The analysis population was participants of all ages with newly-diagnosed high-grade CIN and lesional tissue samples analyzed for HPV types
Measure: Number; unit: Cases per 100,000 women
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 289 | 311 | 285 | 299 | 390 | 304
Cases per 100,000 women
  Overall CIN | 164.2 [0.6 to 4.0] | 230.9 [0.0 to 1.8] | 133.3 [0.0 to 1.9] | 149.6 [0.0 to 1.8] | 142.6 [0.3 to 2.6] | 200.3 [0.2 to 2.9]
  HPV 6/11/16/18-related CIN | 80.6 | 115.0 | 70.1 | 75.1 | 73.9 | 106.2

11. Primary Outcome: Incidence of HPV 6/11/16/18-related Cervical Intraepithelial Neoplasia for Participants <=26 Years of Age
Description: as for outcome 10
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: The analysis population was participants <=26 years of age with newly-diagnosed high-grade CIN and lesional tissue samples analyzed for HPV types
Measure: Number; unit: Cases per 100,000 women
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 74 | 100 | 42 | 33 | 103 | 93
Cases per 100,000 women
  Overall CIN | 133.4 [0.6 to 4.0] | 198.6 [0.0 to 1.8] | 71.3 [0.0 to 1.9] | 76.1 [0.0 to 1.8] | 94.1 [0.3 to 2.6] | 156.8 [0.2 to 2.9]
  HPV 6/11/16/18-related CIN | 72.2 | 117.2 | 50.9 | 41.6 | 56.6 | 102.9

12. Primary Outcome: Incidence of HPV 6/11/16/18-related Cervical Intraepithelial Neoplasia for Participants >26 Years of Age
Description: as for outcome 10
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: The analysis population was participants >26 years of age with newly-diagnosed high-grade CIN and lesional tissue samples analyzed for HPV types
Measure: Number; unit: Cases per 100,000 women
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 215 | 211 | 243 | 266 | 287 | 211
Cases per 100,000 women
  Overall CIN | 179.5 [0.6 to 4.0] | 251.3 [0.0 to 1.8] | 172.6 [0.0 to 1.9] | 196.2 [0.0 to 1.8] | 140.8 [0.3 to 2.6] | 228.3 [0.2 to 2.9]
  HPV 6/11/16/18-related CIN | 85.1 | 114.3 | 85.3 | 97.3 | 68.7 | 108.2

13. Primary Outcome: Incidence of Cervical Intraepithelial Neoplasia Associated With High-risk HPV Types Other Than 16/18 in Participants <=26 Years of Age
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. In addition, lesional tissue samples were routinely collected and stored; the 2004 to 2006 period was chosen because it was sufficiently recent to reflect HPV type status immediately before licensure of Gardasil. The percentage of new cases of high-grade (2/3) CIN related to high-risk HPV types other than 16 and 18 was analyzed. High-risk HPV types include 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, and 68. Incidence was age-adjusted according to Nordic Standard Population.
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: as for outcome 11
Measure: Number; unit: Cases per 100,000 women
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 74 | 100 | 42 | 33 | 103 | 93
Cases per 100,000 women
  Overall CIN | 133.4 [30.8 to 42.3] | 198.6 [32.5 to 43.6] | 71.3 [26.6 to 37.7] | 76.1 [30.7 to 41.8] | 94.1 [32.1 to 41.9] | 156.8 [29.8 to 40.9]
  CIN not related to HPV 16/18 | 46.8 | 67.5 | 17.0 | 30.0 | 34.7 | 45.5

14. Primary Outcome: Incidence of Cervical Intraepithelial Neoplasia Associated With High-risk HPV Types Other Than 16/18 in Participants >26 Years of Age
Description: as for outcome 13
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: as for outcome 12
Measure: Number; unit: Cases per 100,000 women
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 215 | 211 | 243 | 266 | 287 | 211
Cases per 100,000 women
  Overall CIN | 179.5 [30.8 to 42.3] | 251.3 [32.5 to 43.6] | 172.6 [26.6 to 37.7] | 196.2 [30.7 to 41.8] | 140.8 [32.1 to 41.9] | 228.3 [29.8 to 40.9]
  CIN not related to HPV 16/18 | 65.9 | 100.0 | 57.5 | 70.0 | 52.0 | 86.5

15. Primary Outcome: Incidence of HPV 6/11/16/18-related Cervical Cancer in Participants of All Ages
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. In addition, lesional tissue samples were routinely collected and stored; the 2004 to 2006 period was chosen because it was sufficiently recent to reflect HPV type status immediately before licensure of Gardasil. The number of new cases of HPV 6/11/16/18-related cervical cancer was estimated based on the proportion of HPV 6/11/16/18 in all cervical cancers in a representative sample. Incidence was age-adjusted according to Nordic Standard Population.
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: The analysis population was participants with newly-diagnosed cervical cancer and lesional tissue samples analyzed for HPV types
Measure: Number; unit: Cases per 100,000 women
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 202 | 203 | 187 | 185 | 148 | 126
Cases per 100,000 women
  Overall cervical cancer | 13.8 [0.6 to 4.0] | 12.4 [0.0 to 1.8] | 11.7 [0.0 to 1.9] | 11.7 [0.0 to 1.8] | 8.4 [0.3 to 2.6] | 8.7 [0.2 to 2.9]
  HPV 6/11/16/18-related cervical cancer | 9.0 | 9.0 | 7.4 | 7.7 | 5.2 | 6.3

16. Primary Outcome: Incidence of HPV 6/11/16/18-related Cervical Cancer in Participants <=26 Years of Age
Description: as for outcome 15
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: The analysis population was participants <=26 years of age with newly-diagnosed cervical cancer and lesional tissue samples analyzed for HPV types
Measure: Number; unit: Cases per 100,000 women
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 9 | 11 | 4 | 5 | 6 | 8
Cases per 100,000 women
  Overall cervical cancer | 2.6 [0.6 to 4.0] | 1.7 [0.0 to 1.8] | 0.9 [0.0 to 1.9] | 1.4 [0.0 to 1.8] | 0.8 [0.3 to 2.6] | 1.0 [0.2 to 2.9]
  HPV 6/11/16/18-related cervical cancer | 2.3 | 1.7 | 0.9 | 1.4 | 0.5 | 0.75

17. Primary Outcome: Incidence of HPV 6/11/16/18-related Cervical Cancer in Participants >26 Years of Age
Description: as for outcome 15
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: The analysis population was participants >26 years of age with newly-diagnosed cervical cancer and lesional tissue samples analyzed for HPV types
Measure: Number; unit: Cases per 100,000 women
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 193 | 192 | 183 | 180 | 142 | 118
Cases per 100,000 women
  Overall cervical cancer | 19.3 [0.6 to 4.0] | 19.2 [0.0 to 1.8] | 18.6 [0.0 to 1.9] | 18.2 [0.0 to 1.8] | 13.3 [0.3 to 2.6] | 13.6 [0.2 to 2.9]
  HPV 6/11/16/18-related cervical cancer | 12.3 | 13.6 | 11.7 | 11.8 | 8.2 | 9.8

18. Primary Outcome: Incidence of Cervical Cancer Associated With High-risk HPV Types Other Than 16/18 in Participants <=26 Years of Age
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. In addition, lesional tissue samples were routinely collected and stored; the 2004 to 2006 period was chosen because it was sufficiently recent to reflect HPV type status immediately before licensure of Gardasil. The percentage of new cases of cervical cancer associated with high-risk HPV types other than 16 and 18 was estimated based on the proportion of HPV 16/18 in all cervical cancer in a representative sample. Incidence was age-adjusted according to Nordic Standard Population.
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: as for outcome 16
Measure: Number; unit: Cases per 100,000 women
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 9 | 11 | 4 | 5 | 6 | 8
Cases per 100,000 women
  Overall cervical cancer | 2.6 [30.8 to 42.3] | 1.7 [32.5 to 43.6] | 0.9 [26.6 to 37.7] | 1.4 [30.7 to 41.8] | 0.8 [32.1 to 41.9] | 1.0 [29.8 to 40.9]
  Cervical cancer not related to HPV 16/18 | 0.3 | 0.0 | 0.0 | 0.0 | 0.1 | 0.0

19. Primary Outcome: Incidence of Cervical Cancer Associated With High-risk HPV Types Other Than 16/18 in Participants >26 Years of Age
Description: as for outcome 18
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: as for outcome 17
Measure: Number; unit: Cases per 100,000 women
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 193 | 192 | 183 | 180 | 142 | 118
Cases per 100,000 women
  Overall cervical cancer | 19.3 [0.6 to 4.0] | 19.2 [0.0 to 1.8] | 18.6 [0.0 to 1.9] | 18.2 [0.0 to 1.8] | 13.3 [0.3 to 2.6] | 13.6 [0.2 to 2.9]
  Cervical cancer not related to HPV 16/18 | 4.6 | 3.6 | 3.5 | 3.4 | 2.8 | 2.0

20. Primary Outcome: Incidence of HPV-related Histologically Confirmed Female Genital Diseases, Including Vulvar and Vaginal Cancer and Their High-grade Precursors
Description: The incidence of HPV-related histologically confirmed female genital diseases, including vulvar and vaginal cancer and their high-grade precursors was to be assessed.
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: Analysis of this endpoint was not planned nor were the data collected. Thus, the number of participants analyzed is zero.
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

21. Primary Outcome: Prevalence of HPV 6/11/16/18 Infection in Participants <=26 Years of Age
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. In addition, lesional tissue samples were routinely collected and stored; the 2004 to 2006 period was chosen because it was sufficiently recent to reflect HPV type status immediately before licensure of Gardasil. The percentage of liquid-based cervical cytology samples positive for HPV 6, 11, 16, or 18 was analyzed.
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: The analysis population was participants <=26 years of age with liquid-based cytology samples analyzed for HPV types
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 831 | 1043 | 1055 | 1011 | 968 | 996
Percentage of participants | 20.3 [17.6 to 23.2] | 14.2 [12.1 to 16.5] | 26.7 [24.1 to 29.5] | 22.6 [20.0 to 25.3] | 19.0 [16.6 to 21.6] | 13.4 [11.3 to 15.6]

22. Primary Outcome: Prevalence of HPV 6/11/16/18 Infection in Participants >26 Years of Age
Description: as for outcome 21
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: The analysis population was participants >26 years of age with liquid-based cytology samples analyzed for HPV types
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 1486 | 1026 | 958 | 1217 | 1196 | 1006
Percentage of participants | 6.3 [5.1 to 7.6] | 4.7 [3.5 to 6.2] | 5.5 [4.2 to 7.2] | 6.2 [4.9 to 7.7] | 5.6 [4.4 to 7.1] | 7.7 [6.1 to 9.5]

23. Primary Outcome: Prevalence of HPV Infection for High-risk Types Other Than 16/18 for Participants <=26 Years of Age
Description: All Nordic countries participating in this study have national cervical cancer screening programs and registry systems that routinely collect information on cervical cytology, histology, and/or definitive therapy results. In addition, lesional tissue samples were routinely collected and stored; the 2004 to 2006 period was chosen because it was sufficiently recent to reflect HPV type status immediately before licensure of Gardasil. The percentage of liquid-based cervical cytology samples positive for high-risk HPV Types other than 16 or 18, and not co-infected with Types 16 or 18, was analyzed.
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: The analysis population was participants <=26 years of age with liquid-based cytology samples analyzed for HPV types
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 831 | 1043 | 1055 | 1011 | 968 | 996
Percentage of participants | 25.6 [22.7 to 28.7] | 22.8 [20.3 to 25.5] | 27.5 [24.8 to 30.3] | 23.5 [21.0 to 26.3] | 21.2 [18.6 to 23.9] | 24.6 [22.0 to 27.4]

24. Primary Outcome: Prevalence of HPV Infection for High-risk Types Other Than 16/18 for Participants >26 Years of Age
Description: as for outcome 23
Time Frame: Three years before Gardasil licensure (2004 to 2006) and two years after Gardasil licensure (2011 to 2012)
Population: The analysis population was participants >26 years of age with liquid-based cytology samples analyzed for HPV types
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Denmark Participants 2004 to 2006 Before Gardasil Licensure | Denmark Participants 2011 to 2012 After Gardasil Licensure | Norway Participants 2004 to 2006 Before Gardasil Licensure | Norway Participants 2011 to 2012 After Gardasil Licensure | Sweden Participants 2004 to 2006 Before Gardasil Licensure | Sweden Participants 2011 to 2012 After Gardasil Licensure
Number analyzed (Participants) | 1486 | 1026 | 958 | 1217 | 1196 | 1006
Percentage of participants | 12.6 [10.9 to 14.4] | 9.0 [7.3 to 10.9] | 9.6 [7.8 to 11.6] | 9.1 [7.6 to 10.9] | 9.0 [7.5 to 10.8] | 11.0 [9.2 to 13.1]

25. Primary Outcome: Percentage of Live Born Babies With a Major Congenital Anomaly
Description: The percentage of live born babies with major congenital anomalies (MCA) born to women vaccinated with Gardasil during pregnancy and to women in the general population was assessed. For Denmark and Sweden diagnoses of congenital anomaly within 1 year of birth are included; for Norway diagnoses at birth are included.
Time Frame: Up to 5 years after Gardasil licensure (2007 to 2011)
Population: The analysis population represents the babies born to participating mothers, instead of female participants, because the number of babies represents the denominator for the percentage calculation, not female participants (i.e., mothers)
Measure: Number; unit: Percentage of babies with a MCA
Groups:
- Babies Born to Denmark Participants Who Received Gardasil: Live babies born between 2007 and 2011 to Denmark participants who received Gardasil during pregnancy
- Babies Born to Denmark Participants: Live babies born between 2007 and 2011 to Denmark participants in the general population, including participants who did and did not receive Gardasil
- Babies Born to Norway Participants Who Received Gardasil: Live babies born between 2007 and 2011 to Norway participants who received Gardasil during pregnancy
- Babies Born to Norway Participants: Live babies born between 2007 and 2011 to Norway participants in the general population, including participants who did and did not receive Gardasil
- Babies Born to Sweden Participants Who Received Gardasil: Live babies born between 2007 and 2011 to Sweden participants who received Gardasil during pregnancy
- Babies Born to Sweden Participants: Live babies born between 2007 and 2011 to Sweden participants in the general population, including participants who did and did not received Gardasil
Arm/Group | Babies Born to Denmark Participants Who Received Gardasil | Babies Born to Denmark Participants | Babies Born to Norway Participants Who Received Gardasil | Babies Born to Norway Participants | Babies Born to Sweden Participants Who Received Gardasil | Babies Born to Sweden Participants
Number analyzed (Participants) | 371 | 320891 | 23 | 306290 | 105 | 543738
Percentage of babies with a MCA | 5.9 | 4.4 | 4.3 | 2.9 | 2.9 | 3.0
Statistical Analysis 1: Comparison: Babies Born to Denmark Participants Who Received Gardasil vs Babies Born to Denmark Participants; Test type: Superiority or Other; Standardized Prevalence Ratio (SPR) = 1.34, 95% CI 2-sided [0.89 to 2.00] — SPR is the age-adjusted ratio of percentage of live births with a major congenital anomaly (Women who received Gardasil / Women in the general population)
Statistical Analysis 2: Comparison: Babies Born to Norway Participants Who Received Gardasil vs Babies Born to Norway Participants; Test type: Superiority or Other; Standardized Prevalence Ratio (SPR) = 1.59, 95% CI 2-sided [0.00 to 4.77] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Babies Born to Sweden Participants Who Received Gardasil vs Babies Born to Sweden Participants; Test type: Superiority or Other; Standardized Prevalence Ratio (SPR) = 0.86, 95% CI 2-sided [0.00 to 2.02] — [estimate comment as in outcome 25, analysis 1]

26. Secondary Outcome: Incidence of Cervical Intraepithelial Neoplasia by Gardasil Vaccination Status
Description: The incidence of CIN by Gardasil vaccination status was to be assessed.
Time Frame: Four years to 5 years after Gardasil licensure (2011 to 2012)
Population: The analysis population was to be women who underwent cervical screening. A joint decision was made by the study team to forgo the stratified analysis by vaccination status because there were few women who had both been vaccinated with Gardasil and undergone cervical cancer screening. Thus, the number of participants analyzed is zero.
Groups:
- Denmark Participants Who Received Gardasil: Denmark participants who received Gardasil on or before March 2012
- Norway Participants Who Received Gardasil: Norway participants who received Gardasil on or before March 2012
- Sweden Participants Who Received Gardasil: Sweden participants who received Gardasil on or before March 2012
Arm/Group | Denmark Participants Who Received Gardasil | Denmark Participants Who Did Not Receive Gardasil | Norway Participants Who Received Gardasil | Norway Participants Who Did Not Receive Gardasil | Sweden Participants Who Received Gardasil | Sweden Participants Who Did Not Receive Gardasil
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Incidence of Cervical Cancer by Gardasil Vaccination Status
Description: The incidence of other cervical cancers by Gardasil vaccination status was to be assessed.
Time Frame: Four years to 5 years after Gardasil licensure (2011 to 2012)
Population: as for outcome 26
Arm/Group | Denmark Participants Who Received Gardasil | Denmark Participants Who Did Not Receive Gardasil | Norway Participants Who Received Gardasil | Norway Participants Who Did Not Receive Gardasil | Sweden Participants Who Received Gardasil | Sweden Participants Who Did Not Receive Gardasil
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Incidence of Other HPV-related Genital Diseases by Gardasil Vaccination Status
Description: The incidence of other HPV-related genital diseases, including vulvar and vaginal cancers, by Gardasil vaccination status was to be assessed.
Time Frame: Four years to 5 years after Gardasil licensure (2011 to 2012)
Population: as for outcome 26
Arm/Group | Denmark Participants Who Received Gardasil | Denmark Participants Who Did Not Receive Gardasil | Norway Participants Who Received Gardasil | Norway Participants Who Did Not Receive Gardasil | Sweden Participants Who Received Gardasil | Sweden Participants Who Did Not Receive Gardasil
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Prevalence of HPV 6, 11, 16, and 18 Infection by Gardasil Vaccination Status
Description: The percentage of participants with liquid-based cervical cytology samples positive for HPV 6, 11, 16, and 18 was to be analyzed by Gardasil vaccination status.
Time Frame: Four years to 5 years after Gardasil licensure (2011 to 2012)
Population: as for outcome 26
Arm/Group | Denmark Participants Who Received Gardasil | Denmark Participants Who Did Not Receive Gardasil | Norway Participants Who Received Gardasil | Norway Participants Who Did Not Receive Gardasil | Sweden Participants Who Received Gardasil | Sweden Participants Who Did Not Receive Gardasil
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Per protocol, adverse events were not collected as part of the study database; therefore, none were collected and the number at risk is zero
Groups:
- Denmark Participants: All Denmark study participants
- Norway Participants: All Norway study participants
- Sweden Participants: All Sweden study participants
Arm/Group | Denmark Participants | Norway Participants | Sweden Participants
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.